CLINICAL TRIAL: NCT00433069
Title: A Pilot Study of Treatment With Pegylated Interferon-Alpha2a, Ribavirin and Insulin Sensitizer Pioglitazone of Insulin Resistance (With the Exception of Diabetes) in Hepatitis C Virus Infection (The INSPIRED HCV Study)
Brief Title: Retreatment of Chronic Hepatitis C Non-responders With Pegylated Interferon Alpha Plus Ribavirin Plus Pioglitazone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Negro Francesco, Professor, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GE-DMI-05-116
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Insulin resistance; Pioglitazone; Non-responders
MeSH Terms: conditions — Hepatitis C, Chronic; Insulin Resistance | interventions — Pioglitazone; Interferon alpha-2; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Pioglitazone 15 mg QD + pegylated interferon Alfa-2a 180 μg QW + ribavirin 1000-1200 mg QD for 12 weeks, to be continued to a total of 48 weeks in case of complete early virological response, defined as undetectable serum HCV RNA after 12 weeks of triple therapy
  Interventions: Drug: Pioglitazone; Drug: Interferon Alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pioglitazone — Increase early virological response to pegylated interferon alpha plus ribavirin by increasing insulin sensitivity
  Other Names: Actos
Drug: Interferon Alfa-2a — Standard of care for chronic hepatitis C
  Other Names: Pegasys
Drug: Ribavirin — Standard of care for chronic hepatitis C
  Other Names: Copegus

SUMMARY:
The aim of this study is to investigate the efficacy and safety of an insulin-sensitizer (Actos) added to a standard Pegasys/Copegus combination therapy of chronic hepatitis C in patients who have previously failed a pegylated-interferon-alpha / ribavirin combination without the insulin sensitizer. The primary endpoint is the initial virological response (level of HCV RNA in serum) as evaluated after 12 weeks of triple therapy.

DETAILED DESCRIPTION:
Insulin resistance and diabetes are major disease modifiers in chronic hepatitis C, as they increase liver fibrogenesis and reduce the rate of response to antivirals. Regarding the latter, a previous study showed that a sustained virological response (SVR) occurred in about one third of patients with genotype 1 and insulin resistance (measured as homeostasis assessment of insulin resistance, HOMA-IR > 2) vs. two thirds of genotype 1 patients without insulin resistance. These findings were independently confirmed by other studies and extended to non-responders with genotypes 2, 3 and 4. Thus, we suggested that insulin resistance should be corrected in patients with chronic hepatitis C not responding to currently available antiviral treatment, in order to improve response to retreatment. The modalities of this intervention, however, have not been established. In addition, the optimal HOMA-IR score to be attained has not been identified. To assess this point, we planned a prospective, multicenter study to investigate the efficacy and safety of the insulin-sensitizer pioglitazone (ActosTM, Takeda Pharma AG, Lachen, Switzerland) 15 mg QD, added to the pegylated interferon-α2a (PEG-IFN-α2a) (PegasysTM, Roche Pharma Schweiz AG, Reinach, Switzerland) 180 μg QW/ribavirin (CopegusTM, Roche) 1000-1200 mg QD combination therapy in chronic hepatitis C patients who had previously failed to respond (i.e. had detectable serum HCV RNA after 12 weeks of therapy) to a pegylated interferon-α/ribavirin combination without the insulin-sensitizer. All patients had a baseline HOMA-IR score >2 as additional inclusion criterion, because this was the threshold discriminating responders from non-responders in previous works. Diabetic patients were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chronic hepatitis C as per liver biopsy performed during the 12 months prior to enrollment (except patients with histologically proven cirrhosis or a Actitest/Fibrotest assay, or a Fibroscan performed during the 12 months prior to enrollment)
* HCV RNA in serum >600 IU/ml
* elevated ALT
* HCV genotypes 1, 2, 3 or 4
* failure to respond to a prior treatment with a pegylated interferon alpha + ribavirin
* HOMA score > 2.00
* documentation that sexually active female patients of childbearing potential are practicing adequate contraception (intrauterine device, oral contraceptives, progesterone implanted rods, medroxyprogesterone acetate, surgical sterilization plus a barrier method [diaphragm + spermicide] or monogamous relationship with a male partner who has had a vasectomy or is using a condom + spermicide) during the treatment period and for 6 months after discontinuation of therapy. A serum pregnancy test obtained at entry prior to the initiation of treatment must be negative. Female patients must not be breast feeding
* documentation that sexually active male patients are practicing acceptable methods of contraception (vasectomy, use of a condom + spermicide, monogamous relationship with a female partner who practices an acceptable method of contraception) during the treatment period and for 6 months after discontinuation of therapy
* willingness and capability to give written informed consent and to comply with the requirements of the trial

Exclusion Criteria:

* history of diabetes (ADA definition)
* history of significant cardiovascular disease (NYHA III) including but not limited to uncontrolled hypertension, angina pectoris, myocardial infarction, coronary artery surgery and congestive heart failure
* HBsAg and/or HIV
* auto-immune disease, including auto-immune hepatitis
* alcohol consumption exceeding 40 grams per day
* hepatocellular carcinoma
* renal insufficiency (serum creatinine levels above 200 micromol/l)
* unconjugated bilirubin blood level > 100 micromol/l
* glutamyl transferase > 20 times the ULN
* prothrombin time < 60% of control (except in case of oral anti-coagulant therapy)
* neutrophil count < 1.5 G/L
* platelet count < 70 G/L
* hemoglobin <120 g/L
* organ or bone marrow transplantation
* current neoplasm and/or anti-tumor chemotherapy
* current hepatic arterial thrombosis
* pregnant or breast feeding women; child bearing potential women without adequate contraception throughout the course of therapy
* psychosis or anti-depressant therapy for uncontrolled clinical depression
* epilepsy
* clinically significant retinal abnormalities
* thyroid dysfunction
* drug abuse or substitution therapy during the 12 months prior to inclusion
* interstitial pneumonitis
* previous auto-immune hemolysis and all causes of chronic hemolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Early virological response | Week 12 of triple combined therapy

SECONDARY OUTCOMES:
Undetectable serum HCV RNA after 4, 24 weeks and 48 weeks of therapy | Week 2, 24 and 48 of therapy
Changes (vs. baseline) of body weight, HOMA score, after 4, 12 and 48 weeks of therapy and after 24 weeks of follow-up | Weeks 4, 12 and 48 of therapy
Improvement (vs. baseline) of glucose tolerance parameters after 12 and 48 weeks of therapy and after 24 weeks of follow-up | Weeks 12 and 48 of therapy; week 24 of FU

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Negro, Prof, Principal Investigator — University of Geneva, Switzerland
Locations (1):
- Service de Gastroentérologie et d'Hépatologie, University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] Romero-Gomez M, Del Mar Viloria M, Andrade RJ, Salmeron J, Diago M, Fernandez-Rodriguez CM, Corpas R, Cruz M, Grande L, Vazquez L, Munoz-De-Rueda P, Lopez-Serrano P, Gila A, Gutierrez ML, Perez C, Ruiz-Extremera A, Suarez E, Castillo J. Insulin resistance impairs sustained response rate to peginterferon plus ribavirin in chronic hepatitis C patients. Gastroenterology. 2005 Mar;128(3):636-41. doi: 10.1053/j.gastro.2004.12.049. PMID 15765399